CLINICAL TRIAL: NCT00366470
Title: A Double Blind, Randomized, Parallel, Placebo Control Design Study to Determine the Effect of Addition of Vitamin D to Conventional Anti TB Therapy
Brief Title: A Clinical Trial to Study the Effect of the Addition of Vitamin D to Conventional Treatment in New Pulmonary Tuberculosis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peter Daley (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor-Investigator, Peter Daley, Lecturer, Christian Medical College, Vellore, India
Organization: Christian Medical College, Vellore, India (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TB-VitaminD; CTRI/2007/091/000008 (Registry Identifier: Clinical Trials Registry of India)
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Vitamin D in doses of 100,000 IU
  Interventions: Drug: A. 100,000 IU Cholecalciferol per dose of 3.3ml
- B (Placebo Comparator)
  Interventions: Other: B. Migliol Oil without Cholecalciferol

INTERVENTIONS:
Drug: A. 100,000 IU Cholecalciferol per dose of 3.3ml — 100,000 IU Cholecalciferol in 3.3ml Migliol (Carrier) oil, once every two weeks for 2 Months
  Arms: A
Other: B. Migliol Oil without Cholecalciferol — 3.3 ml Migliol Oil, every two weeks for two months
  Arms: B

SUMMARY:
There is some evidence that supplemental Vitamin D may contribute to quicker recovery from TB when given in addition to normal TB therapy. This needs to be proven with a controlled clinical trial. People receiving Vitamin D with anti TB therapy will be compared against people receiving anti TB therapy alone to see if vitamin D contributes to a quicker recovery (as shown by a quicker sputum culture conversion).

DETAILED DESCRIPTION:
The proposed study is a parallel, randomized, double-blinded, placebo-controlled clinical trial to quantify the change, if any, in microbiological outcome in TB patients treated with vitamin D in combination with standard DOTS therapy. It will take place in four South Indian DOTS centres. The required sample size is 250 patients receiving ATT, to be randomised in a 1:1 fashion (125 patients to receive vitamin D and 125 patients to receive placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed smear positive pulmonary tuberculosis.
2. Age between 18 to 75 years
3. No pre-existing liver or renal disease
4. Available for return visits as outlined in the trial protocol
5. A Firm home address

Exclusion Criteria:

1. Extra-pulmonary or smear negative tuberculosis
2. Patients receiving steroids, cytotoxic drugs, post transplant or metastatic malignancy, or not expected to survive for the duration of ATT
3. Pregnant or lactating women
4. Active diarrhoea, indicating possible fat-soluble vitamin malabsorption.
5. Baseline Hypercalcemia >10.5 mg/dl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Time to sputum culture conversion | 8 weeks of treatment

SECONDARY OUTCOMES:
Percent of Patients Culture Positive | 8 Weeks
Performance Status | 8 Weeks
Time To Sputum Smear Conversion | Continous
Proportion of Patients Smear Positive | 4 Weeks, 8 Weeks, 12 Weeks
Time To Growth In Liquid Media | 8 Weeks
RNTCP Treatment Outcomes | 24 Weeks
Weight Gain | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dilip Mathai, MD, FCAMS, Principal Investigator — Christian Medical College, Vellore, India
Locations (2):
- India (2):
  - Bethesda Hospital, Ambur, Tamil Nadu
  - Christian Medical College, Vellore, Tamil Nadu

REFERENCES:
- [Derived] Daley P, Jagannathan V, John KR, Sarojini J, Latha A, Vieth R, Suzana S, Jeyaseelan L, Christopher DJ, Smieja M, Mathai D. Adjunctive vitamin D for treatment of active tuberculosis in India: a randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2015 May;15(5):528-34. doi: 10.1016/S1473-3099(15)70053-8. Epub 2015 Apr 8. PMID 25863562
- See also: TB control in India — http://www.tbcindia.org/pdfs/TB%20India-2005%20Page%201-54.pdf